CLINICAL TRIAL: NCT03083522
Title: Efficacy and Safety of Ojeok-san on Korean Patients With Cold Hypersensitivity in the Hands and Feet - A Randomized, Double-blinded, Placebo Controlled, Multi-center Pilot Study
Brief Title: Efficacy and Safety of Ojeok-san on Korean Patients With Cold Hypersensitivity in the Hands and Feet
Acronym: OJS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chan-Yong Jeon (Other)
Collaborators: Kyunghee University Medical Center (Other); Kyung Hee University Hospital at Gangdong (Other); Semyung University Affiliated Oriental Medical Hospital (Other)
Responsible Party: Sponsor-Investigator, Chan-Yong Jeon, PhD, Gachon University Gil Oriental Medical Hospital
Organization: Gachon University Gil Oriental Medical Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISEE_2017_OJS
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Cold Hypersensitivity
Keywords: Cold Hypersensitivity; Korean medicine; Ojeok-san; Cold intolerance
MeSH Terms: conditions — Cold Hypersensitivity | interventions — ojeok-san; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OJS group (Experimental): admission to Ojeok-san granule
  Interventions: Drug: Ojeok-San
- Placebo Group (Placebo Comparator): admission to placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ojeok-San — Usage: 3g, three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Other Names: OJS
  Arms: OJS group
Drug: Placebo — Usage: 3g three times a day, each taken before or between meals Manufacturing company: HANPOONG PHARM & FOODS Co. Ltd.
  Other Names: corn starch
  Arms: Placebo Group

SUMMARY:
The Purpose of this trial is to investigate the efficacy and safety of Ojeok-san(OJS) on Korean Patients With Cold Hypersensitivity in the Hands

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged 19 to 59 years have a complaint of CHH.
2. Patients must include at least one or more of the following symptoms:

   * Those who have the symptoms of CHH in normal temperature which most individuals feel no cold;
   * Those who have the symptoms of extremely cold hands in cold temperature exposure;
   * Those who are on the return to a warmer environment, the symptoms of cold hands is not completely rewarmed;
3. Those who have 4 cm or greater of VAS CHH score;
4. A thermal differences between the palm (PC8) and the upper arm (LU4) may be higher than 0.3℃;
5. Those who can comply with all study-related procedures, medications, and evaluations;
6. Given a written informed consent form.

Exclusion Criteria:

1. Patients with calcium antagonists or beta-blockers with the purpose of treating CHH;
2. Those who have one or more finger gangrene or ulceration;
3. Those who are diagnosed by hypothyroidism or currently medicated to thyroid drugs;
4. Those who are diagnosed by autoimmune disease or have a positive ANA test result;
5. Those who are diagnosed by carpal tunnel syndrome or have a positive Tinel and Phalen's tests;
6. Those who are diagnosed with cervical disc herniation or (malignant) tumor disease;
7. Those who are diagnosed with diabetes;
8. Those who are currently medicated to drugs that may affect to CHH symptoms, such as anticoagulants etc;
9. Those who have moderate level of liver dysfunction (each of AST, ALT greater than 100 IU/L) or kidney dysfunction (Cr 2.0mg/dL);
10. Those who do not (cannot) abide by treatment and follow up due to the mental illness such as behavior disorder, depression, anxiety neurosis, schizophrenia, or serious mental illness;
11. Those who are Diagnosed with moderate anemia and hematologic disorders (adult non-pregnant women hemoglobin (Hgb) level less than 7g/dL, hematocrit (Hct) level less than 26%, white blood cell (WBC) level greater than 11,000/mm3);
12. Those whose systolic blood pressure (SBP) 180mmHg or diastolic blood pressure (DBP) is greater than 100 mmHg based on average value of at least 2 measurements;
13. Those who are suspected arrhythmia that showing up on ECG, or diagnosed by heart diseases, such as, ischemic heart disease and so on;
14. Those who are addicted to alcohol or drugs;
15. Those who are pregnant (positive urine-HCG) or lactating or have the chances of pregnancy;
16. Those who are diagnosed with malignant tumor
17. Those who are currently participated in other clinical trials;
18. Those who are unable to understand and speak Korean;
19. Those who are judged to be inappropriate for the clinical study by the researchers.

Ages: 19 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in visual analogue scale | At baseline, week 4, 8, 12

SECONDARY OUTCOMES:
Changes from baseline in body temperature | At baseline, week 4, 8, 12
Changes from baseline in WHOQoL-BREF | At baseline, week 4, 8, 12
Changes from baseline in cold stress test | At baseline, week 8
  similar to the cold stimulation test
Vital Sign | every visit
  Body temperature, blood pressure, pulse rate
Liver function tests | At screening visit, week 8
  Levels of AST, ALT and r-GTP
Kidney function test | At screening visit, week 8
  Levels of BUN and Cr
complete blood count | At screening visit, week 8
Adverse event | At week 4, 8, 12

OTHER OUTCOMES:
Pattern Identification Questionnaire | At screening visit
  This questionnaire is a traditional medicine researcher self-developed questionnaire for collecting general symptoms of patients with Cold Hypersensitivity in the Hands and feet
Cold Hypersensitivity diagnostic tool | At screening visit
  This tool is a traditional medicine researcher self-developed questionnaire of screening for patients with Cold Hypersensitivity in the Hands and feet In this trial, we will assess the validity of the tool.

CONTACTS AND LOCATIONS:
Overall Officials: Chanyong Jeon, PhD, Study Chair — Gachon University Gil Oriental Medical Hospital
Locations (1):
- Kyung Hee university medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ko Y, Go HY, Han IS, Lee KY, Kim TH, Lee JM, Jang JB, Song YK, Sun SH, Jeon CY, Ko SG. Efficacy and safety of Ojeok-san in Korean female patients with cold hypersensitivity in the hands and feet: study protocol for a randomized, double-blinded, placebo-controlled, multicenter pilot study. Trials. 2018 Nov 29;19(1):662. doi: 10.1186/s13063-018-3013-9. PMID 30497488